CLINICAL TRIAL: NCT00770562
Title: A Randomized, Open-label Study of First-line Treatment With Dexamethasone or Dexamethasone Plus MabThera on Sustained Treatment Response in Adult Patients With Idiopathic Thrombocytopenic Purpura
Brief Title: A Study Evaluating the Addition of MabThera (Rituximab) to Standard Treatment in Patients With Idiopathic Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18542
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Dexamethasone

ARMS (2):
- Dexamethasone (Active Comparator): Participants received 40 milligrams (mg) dexamethasone, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4). Participants in this treatment arm who failed to achieve a sustained response and had a platelet count of less than or equal to (≤)20 x 10^9 platelets per liter (L; from Day 30 up to end of 6 months) were treated with salvage treatment of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg per square meter (mg/m^2), intravenously (IV), with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28.
  Interventions: Drug: Dexamethasone
- Dexamethasone plus Rituximab (Experimental): Participants received dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV, with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28. Nonresponsive participants with platelets less than (<) 20 x10^9/L or with active bleeding could have also received an additional treatment course of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV on Days 7, 14, 21, and 28 administered with immunoglobulin (IgG) IV (at investigator discretion) and/or low/medium dose steroids (at investigator discretion) on Days 7, 14, 21, and 28.
  Interventions: Drug: rituximab; Drug: Dexamethasone

INTERVENTIONS:
Drug: rituximab
  Other Names: MabThera/Rituxan
  Arms: Dexamethasone plus Rituximab
Drug: Dexamethasone

SUMMARY:
This study will compare the efficacy, safety, and pharmacokinetics of standard treatment versus standard treatment plus MabThera in patients with ITP. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* untreated ITP.

Exclusion Criteria:

* ITP with relapse;
* positive test result for HIV or hepatitis B or C;
* active infection requiring systemic therapy;
* malignancy within 3 years before study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (20):
- Italy (20):
  - Bari
  - Bologna
  - Brescia
  - Cagliari
  - Cuneo
  - Genova
  - Milan
  - Napoli
  - Padua
  - Palermo
  - Pavia
  - Pesaro
  - Pescara
  - Ravenna
  - Reggio Emilia
  - Roma
  - Siena
  - Taranto
  - Udine
  - Verona

REFERENCES:
- [Derived] Zaja F, Baccarani M, Mazza P, Bocchia M, Gugliotta L, Zaccaria A, Vianelli N, Defina M, Tieghi A, Amadori S, Campagna S, Ferrara F, Angelucci E, Usala E, Cantoni S, Visani G, Fornaro A, Rizzi R, De Stefano V, Casulli F, Battista ML, Isola M, Soldano F, Gamba E, Fanin R. Dexamethasone plus rituximab yields higher sustained response rates than dexamethasone monotherapy in adults with primary immune thrombocytopenia. Blood. 2010 Apr 8;115(14):2755-62. doi: 10.1182/blood-2009-07-229815. Epub 2010 Feb 3. PMID 20130241

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Dexamethasone: Participants received 40 milligrams (mg) dexamethasone, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4). Participants in this treatment arm who failed to achieve a sustained response and had a platelet count of less than or equal to (≤)20 x 10^9 platelets per liter (L; from Day 30 up to end of 6 months) were treated with salvage treatment of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg per square meter (mg/m^2), intravenously (IV), with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28.
- Arm B: Dexamethasone + Rituximab: Participants received dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV, with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28. Nonresponsive participants with platelets less than (<) 20 x10^9/L or with active bleeding could have also received an additional treatment course of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV on Days 7, 14, 21, and 28 administered with immunoglobulin (IgG) IV (at investigator discretion) and/or low/medium dose steroids (at investigator discretion) on Days 7, 14, 21, and 28.
Period: Overall Study
Arm/Group | Arm A: Dexamethasone | Arm B: Dexamethasone + Rituximab
Started | 53 | 50
Completed | 52 | 49
Not Completed | 1 | 1
Not completed — Did not take treatment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Dexamethasone: Participants received 40 mg dexamethasone, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4). Participants in this treatment arm who failed to achieve a sustained response and had a platelet count of ≤20 x 10^9 platelets per liter (L; from Day 30 up to end of 6 months) were treated with salvage treatment of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV, with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28.
- Arm B: Dexamethasone + Rituximab: Participants received dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg per square meter (mg/m^2), IV, with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28. Nonresponsive participants with platelets <20 x10^9/L or with active bleeding could have also received an additional treatment course of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV on Days 7, 14, 21, and 28 administered with IgG IV (at investigator discretion) and/or low/medium dose steroids (at investigator discretion) on Days 7, 14, 21, and 28.
- Total: Total of all reporting groups
Arm/Group | Arm A: Dexamethasone | Arm B: Dexamethasone + Rituximab | Total
Number analyzed (Participants) | 52 | 49 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (19) | 49 (16) | 48.41 (18.03)
Sex: Female, Male [Count of Participants; unit: Participants] — Two participants were not accessed because they did not take the study drug after being randomized.
  Participants
    Female | 33 | 27 | 60
    Male | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Sustained Response
Description: Sustained response defined as a platelet count of greater than or equal to (≥) 50x10^9/L at 6 months (Week 24) after the initial treatment. Participants failing therapy before Month 6 (Week 24) and treated in other ways were considered failures.
Time Frame: Week 24
Population: The Intent-to-Treat (ITT) population includes all participants who were randomized, who received at least (<) 1 dose of study medication, and who had at least 1 follow-up contact.
Measure: Number; unit: percentage of participants
Groups:
- Arm A: Dexamethasone: Participants received 40 mg dexamethasone, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4). Participants in this treatment arm who failed to achieve a sustained response and had a platelet count of ≤20 x 10^9/L (from Day 30 up to end of 6 months) were treated with salvage treatment of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV, with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28.
- Arm B: Dexamethasone + Rituximab: Participants received dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV, with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28. Nonresponsive participants with platelets <20 x10^9/L or with active bleeding could have also received an additional treatment course of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV on Days 7, 14, 21, and 28 administered with IgG IV (at investigator discretion) and/or low/medium dose steroids (at investigator discretion) on Days 7, 14, 21, and 28.
Arm/Group | Arm A: Dexamethasone | Arm B: Dexamethasone + Rituximab
Number analyzed (Participants) | 52 | 49
percentage of participants | 36 | 63
Statistical Analysis 1: Comparison: Arm A: Dexamethasone vs Arm B: Dexamethasone + Rituximab; Test type: Superiority or Other; p = 0.004, Fisher Exact

2. Secondary Outcome: Percentage of Participants With an Initial Response
Description: Initial response was defined as an increase in platelet count of ≥50x10^9/L by Day 30 (Week 4) after the start of treatment in either treatment arm.
Time Frame: Week 4
Population: ITT population; excluding participants who received additional steroid therapy or IV Ig course during the first month of therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Dexamethasone | Arm B: Dexamethasone + Rituximab
Number analyzed (Participants) | 44 | 25
percentage of participants | 27 | 68
Statistical Analysis 1: Comparison: Arm A: Dexamethasone vs Arm B: Dexamethasone + Rituximab; Test type: Superiority or Other; p = 0.001, Fisher Exact

3. Secondary Outcome: Percentage of Participants With an Initial Complete Response
Description: Initial complete response was defined as an increase in platelet count of ≥100x10^9/L by Day 30 (Week 4) after the initiation of treatment in either treatment arm.
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Dexamethasone | Arm B: Dexamethasone + Rituximab
Number analyzed (Participants) | 44 | 25
percentage of participants | 23 | 48
Statistical Analysis 1: Comparison: Arm A: Dexamethasone vs Arm B: Dexamethasone + Rituximab; Test type: Superiority or Other; p = 0.015, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Arm A: Dexamethasone: Participants received 40 mg dexamethasone, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4).
- Arm B: Dexamethasone + Rituximab: Participants received dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV, with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28.
- Salvage Therapy: Nonresponsive (failed to achieve a sustained response) participants from Arm A (dexamethasone monotherapy) who had a platelet count of ≤20 x 10^9/L (from Day 30 up to end of 6 months) were treated with salvage treatment of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV, with premedication of oral acetaminophen 500 mg and chlorpheniramine 10 mg IV on Days 7, 14, 21, and 28. Nonresponsive participants from Arm B (dexamethasone + rituximab) with platelets <20 x10^9/L or with active bleeding were treated with salvage therapy of dexamethasone 40 mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4) and rituximab 375 mg/m^2, IV on Days 7, 14, 21, and 28 administered with IgG IV (at investigator discretion) and/or low/medium dose steroids (at investigator discretion) on Days 7, 14, 21, and 28.
Arm/Group | Arm A: Dexamethasone | Arm B: Dexamethasone + Rituximab | Salvage Therapy
Serious Adverse Events (participants affected / at risk) | 1/52 | 3/49 | 3/27
Other Adverse Events (participants affected / at risk) | 25/52 | 37/49 | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Dexamethasone (N=52) | Arm B: Dexamethasone + Rituximab (N=49) | Salvage Therapy (N=27)
Hemorrhage syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Interstitial pneumonia (Infections and infestations) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
TIA (Nervous system disorders) | 0 | 0 | 1
Hemorrhagic syndrome and low platelet (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Dexamethasone (N=52) | Arm B: Dexamethasone + Rituximab (N=49) | Salvage Therapy (N=27)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 7 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 2 | 5 | 0
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 0
Gravitational oedema (General disorders) | 0 | 1 | 0
Hyperpyrexia (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Mucosal hyperaemia (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 10 | 5
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Bronchitis acute (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Helicobacter infection (Infections and infestations) | 1 | 2 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 2 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 4 | 0
Pharyngitis (Infections and infestations) | 1 | 2 | 0
Tinea versicolour (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 2
Tracheitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood amylase increased (Investigations) | 0 | 1 | 0
Blood pressure abnormal (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 0 | 2
Transaminases increased (Investigations) | 3 | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 3 | 6 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Strangury (Renal and urinary disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1
Phlebitis superficial (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights